# Delving Into Borderline Personality Disorder Clinical Trials - Uncovering Clinical Trial Engagement Among Individuals with Borderline Personality Disorder

The Informed Consent Process in <u>Power Clinical Trial's</u>
Observational Study: A Guide for Participants With Borderline
Personality Disorder

Date: August 4, 2023

### This Informed Consent Form Explained

Should you find yourself tasked with filling out this form, it indicates that you are being considered for participation in an observational clinical trial that squarely addresses individuals grappling with borderline personality disorder. The form serves as a detailed guide, unveiling the study's overarching aims, the meticulous plan of execution, and the multifaceted implications, both positive and otherwise. Undertaking a thoughtful contemplation of your potential involvement before reaching a decision is vital, and leaning on the counsel of a trusted confidant can offer valuable insights. If any nuances of the information encapsulated within this document remain shrouded or if queries emerge, rest assured that the researcher stands prepared to provide clarifications.

## Purpose of the Study

Borderline Personality Disorder (BPD) is a mental health condition characterized by a pervasive pattern of instability in relationships, self-image, emotions, and behavior. Individuals with BPD often struggle with intense mood swings, impulsivity, difficulties in forming and maintaining relationships, and a deep fear of abandonment.

People with BPD may have a distorted sense of self and experience rapid shifts in their self-identity, values, and goals. They may also engage in risky behaviors such as self-harm, substance abuse, and reckless driving. Additionally, intense and unstable emotions can lead to anger, depression, and anxiety, often triggered by seemingly minor events.

Borderline personality disorder clinical trials serve as crucial endeavors aimed at scrutinizing the safety and effectiveness of novel treatments for this condition. These trials are indispensable in discerning whether these emerging treatments surpass their existing counterparts and in providing substantiated evidence to endorse their application within the broader population.

The central focus of this particular study is to meticulously examine the encounters of individuals diagnosed with borderline personality disorder as they actively partake in a distinct clinical trial centered on medical interventions. The primary emphasis lies in meticulously tracing the rates of trial completion and voluntary withdrawal among these participants.

#### Introduction to Observational Studies

As a participant in this medical trial, you will be a part of an observational study, which is a type of clinical trial that aims to gather information by observing individuals without making any changes to their care plans.

Researchers will simply observe you and measure the outcomes of the condition without intervening in any way. This type of trial is an important tool for gaining a deeper understanding of the natural progression of a particular condition, and the effects it has on individuals who are diagnosed with it. By participating in this observational study, you will be contributing to the advancement of medical knowledge and helping to improve the care of individuals who have the same condition.

Comparative Insights into Further Borderline Personality Disorder Clinical Trials

It's essential to acknowledge that this clinical trial adopts an observational approach, indicating that your involvement will not encompass the administration of specific treatments or interventions as a constituent of the study. Nonetheless, the landscape of borderline personality disorder clinical trials encompasses a spectrum of variations,

including interventional trials that necessitate participants to undergo specific treatment protocols.

Formulating a well-informed decision regarding your potential engagement in a clinical trial necessitates a proactive approach to researching and contrasting diverse studies. A wealth of information regarding borderline personality disorder-related studies can be accessed through platforms such as clinicaltrials.gov. Furthermore, Power's dedicated website presents an array of borderline personality disorder clinical trials that are actively seeking participants. By dedicating time to meticulous research and comprehending the diverse array of clinical trial formats, you can confidently arrive at a decision regarding your participation in a trial.

### Voluntary Participation in Clinical Trial Surveys

As a participant in this observational clinical trial, we would like to gather information about your experiences. This will be done through the completion of questionnaires every two weeks, which should take approximately 20-30 minutes. In addition, we will conduct check-in calls on a quarterly basis for as long as you continue to participate in the trial.

It's important to emphasize that your participation in the survey aspect of the trial is completely optional. You are not required to answer any or all questions, and you have the right to terminate your involvement in the trial at any time if you so choose. We understand that participating in a clinical trial can be a personal decision, and we are committed to supporting you in any way we can. Your privacy and comfort are of the utmost importance to us, and we will respect your decision-making process throughout the trial.

# Preserving Confidentiality of Your Responses

Upholding the sanctity of your information remains paramount throughout the course of this clinical trial. In the interest of ensuring your anonymity, we kindly request that you abstain from divulging any personal or identifiable particulars within your questionnaire responses. The dedicated research team is resolute in their commitment to fortify the shield of your confidentiality. Nevertheless, it's prudent to acknowledge that specific legal circumstances may arise, necessitating the disclosure of your data.

#### **Benefits**

While immediate benefits may not be evident for individuals partaking in this observational clinical trial, their involvement carries the potential to etch a lasting imprint on the lives of others. The reservoir of data amassed from participants will fuel the refinement of future borderline personality disorder patient enrollment procedures, culminating in heightened accessibility to medical research avenues. By embarking on this clinical journey, individuals seize the opportunity to become catalysts for transformative change within the realm of medical research, significantly impacting the trajectory of future borderline personality disorder patients.

### Risks

The landscape of clinical trials has undoubtedly propelled medical progress, yet it's equally vital to acknowledge the specter of health risks that can loom over participants, particularly in trials involving novel treatments.

However, our observational clinical trial stands as an exception, effectively negating this risk by abstaining from mandating participants to undertake novel interventions. Instead, the focal point revolves around observation and outcome measurement, sans the imposition of any unwarranted health hazards.

# A Voluntary Choice

The journey into the borderline personality disorder clinical trial unfolds as a tapestry woven with voluntarism. The compass of choice navigates solely by your hand, bestowing upon you the prerogative to take a step into this study or redirect your path. Should the decision steer you toward participation, the formalized connection materializes through your signature on the informed consent form. Importantly, this covenant doesn't seal the door of autonomy; rather, it preserves your freedom to disengage from the journey at any juncture, liberating you from the obligation to furnish a rationale for your choice.

Embarking on a Deeper Exploration of Clinical Trial Inclusiveness

For those who nurture an inclination to delve into the multifaceted domain of representation in clinical trials, an array of online resources awaits your eager engagement.

Whether you seek to decipher the tapestry woven with challenges and opportunities, or simply aspire to enrich your own expedition through the realm of clinical trials, these reservoirs of knowledge stand as beacons of insight:

Khozin, Sean, and Andrea Coravos. "Decentralized trials in the age of real-world evidence and inclusivity in clinical investigations." *Clin Pharmacol Ther* 106, no. 1 (2019): 25-27.

Pepperrell, Toby, Florence Rodgers, Pranav Tandon, Kelly Sarsfield, Molly Pugh-Jones, Theo Rashid, and Sarai Keestra. "Making a COVID-19 vaccine that works for everyone: ensuring equity and inclusivity in clinical trials." *Global Health Action* 14, no. 1 (2021): 1892309.

# **Expression of Informed Consent**

I hereby validate that I have devoted substantial time to thoroughly grasp and assimilate the contents encapsulated within the informed consent form, either autonomously or with the support of a trusted individual who has conveyed its essence to me. All queries and reservations that occupied my thoughts have been diligently addressed to my absolute satisfaction.

I am unequivocally cognizant that my engagement in this study materializes through voluntary choice, and the prerogative to revoke my consent rests solely with me, devoid of any obligation to proffer rationale or incur financial obligations. It has been explicitly conveyed to me that a duplicate of this informed consent form shall be tendered for my archival purposes.

After scrupulously weighing and appraising the entirety of the information presented to me, I extend my concurrence to partake in this study, an embodiment of my independent volition.

| Printed Name of Participant |
|-----------------------------|

| Participant Signature |
|---|
| Date |
| Validation by Informed Consent Facilitator |
| I assertively confirm that I have diligently engaged in an extensive dialogue with the participant, meticulously unraveling the intricacies encapsulated within this textual composition. My objective was to ensure the participant's attainment of a crystal-clear comprehension of the trial's overarching objectives, methodologies employed, potential hazards and benefits, as well as other cardinal elements intrinsic to the borderline personality disorder clinical trial. |
| Adequate space was provided to the participant, fostering the emergence of queries and facilitating the rectification of ambiguities or misconceptions. It is imperative to underscore that the participant's engagement in this trial is an act of unimpeded volition, and they enjoy the unrestricted prerogative to terminate their involvement at any juncture, driven by any rationale, without shouldering any financial encumbrance. |
| Following the participant's provision of consent, a meticulously preserved duplicate of this textual document was conferred upon them, serving as a repository for their individual records. |
| Printed Name of Person Taking Consent |
| Signature of Person Taking Consent |
| Date |